CLINICAL TRIAL: NCT00261183
Title: The Contribution of Melatonin Vs. Placebo in Benzodiazepine Withdrawal in Methadone Maintenance Treatment Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-05-SS-03186-CTIL
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2005-12-02 (Estimated); Status verified 2005-11

CONDITIONS: Benzodiazepines
MeSH Terms: interventions — Melatonin

INTERVENTIONS:
Drug: Melatonin

SUMMARY:
We hypothesized that patient will success in benzodiazepine withdrawal if they get melatonin to solve sleep-problems which commonly occur during benzodiazepine withdrawal. Former heroin addicts, currently in Methadone maintenance treatment, who are also abusing benzodiazepine, started self benzodiazepine withdrawal, and got for 6 weeks melatonin (5mg/day, taken every night) or placebo and after 1 week, additional 6 weeks with placebo or melatonin (double blind for what got first).Success The benzodiazepine withdrawal success was evaluated by urine for benzodiazepines, and sleep quality was evaluated using PSQI questionnaire (baseline,and after weeks 6, 7, 13)

DETAILED DESCRIPTION:
A total of 100 patients will participate. Follow-up of benzodiazepines in urine after study and 6 months later will be evaluated, as well as sleep quality (using PSQI)

ELIGIBILITY:
Inclusion Criteria:

* Former opiates addicts, currently in methadone maintenance treatment, and abusing benzodiazepines who intend to withdrawal
* adults (>=18y)

Exclusion Criteria:

* non abusing benzodiazepine
* Refuse making benzodiazepines withdrawal
* non methadone maintenance treatment patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-12; Study Completion 2006-12

PRIMARY OUTCOMES:
Stop benzodiazepine abuse(Urine)

SECONDARY OUTCOMES:
sleep quality (self report- PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Schreiber, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Shaul Schreiber, Tel Aviv, Israel

REFERENCES:
- [Derived] Possemato K, Johnson EM, Emery JB, Wade M, Acosta MC, Marsch LA, Rosenblum A, Maisto SA. A pilot study comparing peer supported web-based CBT to self-managed web CBT for primary care veterans with PTSD and hazardous alcohol use. Psychiatr Rehabil J. 2019 Sep;42(3):305-313. doi: 10.1037/prj0000334. Epub 2018 Nov 29. PMID 30489140
- [Derived] Peles E, Hetzroni T, Bar-Hamburger R, Adelson M, Schreiber S. Melatonin for perceived sleep disturbances associated with benzodiazepine withdrawal among patients in methadone maintenance treatment: a double-blind randomized clinical trial. Addiction. 2007 Dec;102(12):1947-53. doi: 10.1111/j.1360-0443.2007.02007.x. Epub 2007 Oct 4. PMID 17916225